CLINICAL TRIAL: NCT06973980
Title: The Effect of High-Intensity Interval Training on Cardiometabolic Risk Factors, Body Composition, and Plasma FABP4 Levels in Sedentary Obese Adults.
Brief Title: HIIT in Sedentary Obese Adults: Effects on Metabolic Risk, Body Composition, and FABP4
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Eastern Mediterranean University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: YDIREL
Record Dates: First submitted 2025-04-18; First posted 2025-05-15 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2025-05

CONDITIONS: High-Intensity Interval Training
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise Group (Experimental): High-Intensity Interval Training (HIIT)
  1-minute interval, 1-minute active recovery 5-minute warm-up, 3-minute cool-down at 60% of peak heart rate.
  Weeks 1-2:
  Intensity at 85% of peak heart rate during work, active recovery at 60% of peak heart rate, 4 sets of 1-minute work.
  Weeks 2-7:
  Intensity at 90% of peak heart rate during work, active recovery at 60% of peak heart rate, 6 sets of 1-minute work.
  Weeks 8-12:
  Intensity at 90% of peak heart rate during work, active recovery at 60% of peak heart rate, 8 sets of 1-minute work.
  Interventions: Other: Exercise
- Control Group (No Intervention): No intervention will be applied to the control group.

INTERVENTIONS:
Other: Exercise — The exercises will be applied only to the intervention group for 12 weeks and will be progressively intensified every 4 weeks.
  Arms: Exercise Group

SUMMARY:
It is aimed to investigate the responses of Fatty Acid Binding Protein 4 (FABP4), which has been discovered as a novel biomarker of obesity and metabolic diseases, to regular exercise training.

The aim of this study is to investigate the effects of high-intensity interval training (HIIT) on cardiometabolic risk factors, body composition, and plasma FABP4 levels in sedentary obese adults.

DETAILED DESCRIPTION:
Fatty acid binding proteins are intracellular proteins involved in the transport of fatty acids and are particularly associated with lipolytic activity. These proteins constitute a group of molecules that regulate intracellular lipid responses and are linked to metabolic and inflammatory pathways.

Studies have shown that FABP4 is associated with hypertension, insulin resistance, obesity, and stroke.

Inhibition of FABP4 synthesis has emerged as a promising strategy for the treatment of obesity-related conditions, particularly insulin resistance and diabetes, and it is emphasized that exercise models to suppress FABP4 should be further investigated.

The aim of this study is to investigate the effects of high-intensity interval training (HIIT) on cardiometabolic risk factors, body composition, and plasma FABP4 levels in sedentary obese adults.

Hypotheses:

H01: HIIT has no effect on cardiometabolic risk factors in sedentary obese adults.

H02: HIIT has no effect on body composition in sedentary obese adults. H03: HIIT has no effect on plasma FABP4 levels in sedentary obese adults.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 20 and 35 years,
* BMI between 30 and 35 kg/m²,
* Waist circumference of 90-100 cm for women, 105-110 cm for men,
* Sedentary lifestyle (<600 MET-min/week),
* Referred by a physician (with a statement confirming no contraindication to exercise)."

Exclusion Criteria:

* BMI > 35,
* Pregnancy,
* Cardiovascular Diseases: Individuals with serious cardiovascular issues, such as uncontrolled hypertension, heart failure, coronary artery disease, or a heart attack within the last 6 months, which could pose a risk during exercise.
* Respiratory Diseases: Individuals with chronic respiratory conditions, such as uncontrolled or severe asthma or COPD, who cannot tolerate exercise due to their condition.
* Neurological Disorders: Individuals with neurological issues that limit exercise capacity, such as Parkinson's disease, stroke, or multiple sclerosis.
* Musculoskeletal Issues: Individuals with chronic musculoskeletal problems, particularly knee or hip osteoarthritis, that may increase the risk of pain or injury during exercise.
* Metabolic or Endocrine Disorders: Individuals with uncontrolled metabolic issues, such as diabetes or thyroid disorders, that could cause blood sugar or hormonal fluctuations during exercise.
* Acute Infections or Illness: Individuals with acute infections, fever, or recently undergone surgical procedures.
* Any health condition that may prevent participation in exercise."

Ages: 20 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Estimated)
Dates: Start 2025-03-01 (Actual); Primary Completion 2025-07-01 (Estimated); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
Fatty acid-bling protein 4 | Baseline, week 6 and week 12
  The Human FABP4 (Fatty Acid Binding Protein 4, Adipocyte) ELISA Kit/96T/Feiyuebio will be used to evaluate fatty acid-binding proteins in the biological samples collected from the participants.
Complete Blood Count | Baseline, week 6 and week 12
  used to evaluate overall health and detect a wide range of disorders, including anemia, infection, and many other diseases.
Hemoglobin A1c (HbA1c) | Baseline, week 6 and week 12
  used to measure the average blood glucose levels over the past 2 to 3 months; commonly used in the diagnosis and management of diabetes.
Hematocrit (HCT) | Baseline, week 6 and week 12
  sed to measure the proportion of red blood cells in the blood; helps evaluate conditions such as anemia, dehydration, and other blood disorders.
Low-Density Lipoprotein | Baseline, week 6 and week 12
  used to measure the level of "bad" cholesterol in the blood; high levels are associated with an increased risk of cardiovascular disease.
High-Density Lipoprotein | Baseline, week 6 and week 12
  Used to quantify the concentration of high-density lipoprotein (HDL) cholesterol in the bloodstream; elevated levels of HDL are inversely correlated with the risk of cardiovascular diseases, suggesting a protective effect on heart health.
Triglycerides | Baseline, week 6 and week 12
  used to measure the concentration of triglycerides (a type of fat) in the blood; elevated levels are associated with an increased risk of cardiovascular disease, metabolic syndrome, and other health conditions.
Fasting Blood Glucose (FBG) | Baseline, week 6 and week 12
  used to measure the concentration of glucose in the blood after an overnight fast; elevated levels may indicate impaired glucose metabolism or diabetes mellitus.
Total Cholesterol | Baseline, week 6 and week 12
  used to measure the overall concentration of cholesterol in the blood, including low-density lipoprotein (LDL), high-density lipoprotein (HDL), and very-low-density lipoprotein (VLDL); elevated levels are associated with an increased risk of cardiovascular diseases.

SECONDARY OUTCOMES:
Physical Activity Level Assessment | Baseline, week 6 and week 12
  The International Physical Activity Questionnaire Short Form will be used. A validity and reliability study has been conducted in Turkish, with test-retest reliability determined to be r=0.69. This form is self-administered and consists of seven questions assessing physical activity levels over the 'last seven days.' It provides information on time spent sitting, walking, engaging in moderate-intensity activities, and vigorous-intensity activities. The score is calculated by multiplying the minutes, days, and MET values. For calculations, 8 MET is used for vigorous physical activity, 4 MET for moderate-intensity activity, and 3.3 MET for walking. Since the scale is openly accessible, no usage permission is required.
Physical activity level | Baseline, week 6 and week 12
  1. High Activity Level: Individuals who engage in vigorous-intensity physical activity (≥8 METs) for at least 3 days per week, accumulating a total of at least 1500 MET-minutes/week, or individuals who engage in any combination of physical activities across 7 days, accumulating at least 3000 MET-minutes/week.
  2. Moderate Activity Level: Individuals who perform vigorous-intensity activity for more than 20 minutes on at least 3 days per week, or moderate-intensity activity for more than 30 minutes on at least 5 days per week, or those who accumulate a total of at least 600 MET-minutes/week through any combination of physical activities.
  3. Low Activity (Sedentary) Level: Individuals whose total physical activity is less than 600 MET-minutes/week are considered sedentary. This indicates minimal physical activity, primarily consisting of sitting, light movement, and a generally inactive lifestyle.
Assessment of Aerobic Capacity and Exercise Intensity - used to measure an individual's maximal oxygen uptake (VO2max) and determine the intensity of exercise | Baseline, week 6 and week 12
  The Bruce Treadmill Test protocol will be used to determine aerobic capacity and exercise intensity. Developed by Robert A. Bruce, the Bruce Treadmill Test protocol is widely used today for non-invasive estimation of VO2max. The incline and speed are regularly increased to reach the maximum level that an individual can achieve. The test consists of 9 stages. Prior to the test, participants will receive the necessary information, and their resting blood pressure, heart rate, and oxygen saturation will be measured. At the end of each stage, an ECG measurement will be taken in addition to these measurements, and at the end of the test, all measurements will be repeated. The peak heart rate obtained at the end of the test will be considered the maximal heart rate. Additionally, the peak heart rate obtained will be used to determine the intensity of the exercise protocols.
Anthropometric Measurements | Baseline, week 6 and week 12
  Height (m) will be assessed by tape
Antropometric Measurement | Baseline, week 6 and week 12
  Body weight (kg) will be assessed using a Body Fat Analyzer.
Antropometric Measurement | Baseline, week 6 and week 12
  body mass indeks (kg/m²) will be calculated

CONTACTS AND LOCATIONS:
Overall Officials: YAŞAM DİREL, MSc, Principal Investigator — Eastern Meditterean university
Locations (1):
- Eastern Mediterranean University, Famagusta, Cyprus

IPD SHARING:
Plan to Share IPD: No